CLINICAL TRIAL: NCT05343039
Title: Leveraging Biomarkers and New Technologies to Reduce Self-Injury and Substance Abuse Risk Among Highly Vulnerable Adolescents
Brief Title: Technology Enhanced Adolescent Mental Health (TEAM)
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-11-6898
Record Dates: First submitted 2022-04-11; First posted 2022-04-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Nonsuicidal Self Injury; Alcohol Abuse; Vagus Nerve Stimulation
Keywords: Adolescence; Emotion Regulation
MeSH Terms: conditions — Self-Injurious Behavior; Alcoholism; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants will receive a tVNS device.
  Interventions: Device: Non-invasive Transcutaneous Nerve Stimulation (tVNS)
- Non-Treatment Group (Experimental): Participants will not receive a tVNS device.
  Interventions: Device: No Intervention

INTERVENTIONS:
Device: Non-invasive Transcutaneous Nerve Stimulation (tVNS) — Participants will engage in 25-minute tVNS sessions every day for 30 days.
  Arms: Treatment Group
Device: No Intervention — Participants will not receive any intervention.
  Arms: Non-Treatment Group

SUMMARY:
Adolescent nonsuicidal self-injury (NSSI) and alcohol misuse, alone and especially in combination, portend significant functional impairment in adulthood (e.g., relationship dysfunction, depression, suicidality). Although psychosocial interventions for NSSI and substance use are effective for some, they are also expensive and require highly trained clinicians. Treatment is therefore often unavailable to disadvantaged adolescents and those who live rurally. Thus, lower-cost alternative treatments are needed. We will evaluate the efficacy of noninvasive transcutaneous vagus nerve stimulation (tVNS), an effective treatment for depression, in reducing risk for NSSI and substance misuse among vulnerable adolescents.

DETAILED DESCRIPTION:
The overarching goals of the proposed project are threefold. AIM 1: Evaluate the clinical efficacy of tVNS in reducing NSSI and alcohol misuse among vulnerable adolescents. We hypothesize that self-administered tVNS, delivered in 25-minute sessions, will reduce self-reported NSSI and alcohol use, improve adolescents' self-reported emotion regulation, and yield improvements in sympathetic and parasympathetic nervous system markers of emotion regulation and vulnerability to NSSI and alcohol misuse. AIM 2: Evaluate treatment adherence compared with traditional psychosocial interventions of similar duration. We hypothesize that adolescents will demonstrate greater treatment adherence than observed in traditional psychosocial interventions of similar duration, and rate tVNS as acceptable, unobtrusive, and favorable to face-to-face treatment. AIM 3: Evaluate maltreatment effects on tVNS. We hypothesize that tVNS will be effective for those with histories of maltreatment.

Although rarely used to date among adolescents, tVNS alters neural and emotional responses to sad stimuli, and among adults, reduces suicide risk up to five years later. At present, it is being evaluated as a treatment for alcohol misuse in a NIH-funded clinical trial. This suggests potential for treating NSSI, alcohol misuse, post-traumatic stress symptoms (PTSS), and other disorders of emotion dysregulation. As outlined above, we will test the efficacy of tVNS in altering behavioral, emotional, and autonomic nervous system risk for NSSI and alcohol misuse, evaluate adherence and acceptability of tVNS among adolescents, and determine if maltreatment histories moderate treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Have used alcohol
* Have engaged in ≥ 3 episodes of NSSI in the past 6 months or ≥ 5 lifetime (1 of these 5 must be in the past year)
* Own a smartphone (iPhone or Android)

Exclusion Criteria:

* Autism
* Schizophrenia
* Have a cardiac pacemaker, implanted defibrillator, or implanted or metallic electronic device
* Pregnant or breastfeeding
* Have a history of seizures or epilepsy
* Temperomandibular Joint Disorder
* Bell's Palsy
* Impaired cranial nerve function or facial pain

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Non-suicidal Self Injury and Alcohol Misuse Behaviors at Day 30 | 30 days
  Participants will engage in 25-minute tVNS sessions daily.
Maintenance of Treatment Effects at 3 Months Post Intervention | 3 months
  Participants will be evaluated on the maintenance of any such treatment effects 3 months post intervention.
Change from Baseline in Emotion Regulation at Day 30 | 30 days
  Participants will complete a 2-3 minute survey daily in which they are to report on different feelings and emotions such as happiness, sadness, and anger.

SECONDARY OUTCOMES:
Adherence to tVNS Intervention from Baseline to Day 30 | 30 days
  Adherence of participants' self-administered daily 25-minute tVNS sessions will be measured from participants' tVNS phone app. They will also report on acceptability, obtrusiveness, and favorability of tVNS.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore P Beauchaine, PhD, Principal Investigator — University of Notre Dame; Brooke A Ammerman, PhD, Principal Investigator — University of Notre Dame; Kristin Valentino, PhD, Principal Investigator — University of Notre Dame
Locations (1):
- University of Notre Dame, South Bend, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson ST, Sears P, Ruvuna F, Bunker M, Conway CR, Dougherty DD, Reimherr FW, Schwartz TL, Zajecka JM. A 5-Year Observational Study of Patients With Treatment-Resistant Depression Treated With Vagus Nerve Stimulation or Treatment as Usual: Comparison of Response, Remission, and Suicidality. Am J Psychiatry. 2017 Jul 1;174(7):640-648. doi: 10.1176/appi.ajp.2017.16010034. Epub 2017 Mar 31. PMID 28359201
- [Background] Achenbach, T.M. (1991). Manual for the youth self-report and 1991 profile. Burlington, VT: University of Vermont Department of Psychiatry.
- [Background] American Foundation for Suicide Prevention. (2021). Project 2025: A nationwide initiative to reduce the annual rate of suicide in the U.S. by 20 percent by 2025. Retrieved on 6/23/2021 from https://project2025.afsp.org/
- [Background] Anestis MD, Pennings SM, Lavender JM, Tull MT, Gratz KL. Low distress tolerance as an indirect risk factor for suicidal behavior: considering the explanatory role of non-suicidal self-injury. Compr Psychiatry. 2013 Oct;54(7):996-1002. doi: 10.1016/j.comppsych.2013.04.005. Epub 2013 May 16. PMID 23684548
- [Background] Beauchaine T. Vagal tone, development, and Gray's motivational theory: toward an integrated model of autonomic nervous system functioning in psychopathology. Dev Psychopathol. 2001 Spring;13(2):183-214. doi: 10.1017/s0954579401002012. PMID 11393643
- [Background] Beauchaine TP. Future Directions in Emotion Dysregulation and Youth Psychopathology. J Clin Child Adolesc Psychol. 2015;44(5):875-96. doi: 10.1080/15374416.2015.1038827. Epub 2015 May 27. PMID 26016727
- [Background] Beauchaine TP, Thayer JF. Heart rate variability as a transdiagnostic biomarker of psychopathology. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):338-350. doi: 10.1016/j.ijpsycho.2015.08.004. Epub 2015 Aug 11. PMID 26272488
- [Background] Beauchaine TP, Cicchetti D. Emotion dysregulation and emerging psychopathology: A transdiagnostic, transdisciplinary perspective. Dev Psychopathol. 2019 Aug;31(3):799-804. doi: 10.1017/S0954579419000671. No abstract available. PMID 31290735
- [Background] Beauchaine TP, Hinshaw SP, Bridge JA. Nonsuicidal Self-Injury and Suicidal Behaviors in Girls: The Case for Targeted Prevention in Preadolescence. Clin Psychol Sci. 2019 Jul;7(4):643-667. doi: 10.1177/2167702618818474. Epub 2019 Jan 28. PMID 31485384
- [Background] Beauchaine TP, Bell Z, Knapton E, McDonough-Caplan H, Shader T, Zisner A. Respiratory sinus arrhythmia reactivity across empirically based structural dimensions of psychopathology: A meta-analysis. Psychophysiology. 2019 May;56(5):e13329. doi: 10.1111/psyp.13329. Epub 2019 Jan 23. PMID 30672603
- [Background] Beauchaine TP, Sauder CL, Derbidge CM, Uyeji LL. Self-injuring adolescent girls exhibit insular cortex volumetric abnormalities that are similar to those seen in adults with borderline personality disorder. Dev Psychopathol. 2019 Oct;31(4):1203-1212. doi: 10.1017/S0954579418000822. PMID 30394252
- [Background] Beauchaine, T. P., & Crowell, S. E. (Eds.) (2020). The Oxford handbook of emotion dysregulation. NY: Oxford University Press.
- [Background] Behavioral Tech. (2021). DBT training and certification. Retrieved on 6/23/2021 from https://behavioraltech.org/re sources/faqs/training-faqs/
- [Background] Bell Z, Shader T, Webster-Stratton C, Reid MJ, Beauchaine TP. Improvements in Negative Parenting Mediate Changes in Children's Autonomic Responding Following a Preschool Intervention for ADHD. Clin Psychol Sci. 2018;6(1):134-144. doi: 10.1177/2167702617727559. Epub 2017 Sep 26. PMID 29545976
- [Background] Berman AH, Bergman H, Palmstierna T, Schlyter F. Evaluation of the Drug Use Disorders Identification Test (DUDIT) in criminal justice and detoxification settings and in a Swedish population sample. Eur Addict Res. 2005;11(1):22-31. doi: 10.1159/000081413. PMID 15608468
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Berntson GG, Cacioppo JT, Quigley KS. Autonomic determinism: the modes of autonomic control, the doctrine of autonomic space, and the laws of autonomic constraint. Psychol Rev. 1991 Oct;98(4):459-87. doi: 10.1037/0033-295x.98.4.459. PMID 1660159
- [Background] Bertrand K, Richer I, Brunelle N, Beaudoin I, Lemieux A, Menard JM. Substance abuse treatment for adolescents: how are family factors related to substance use change? J Psychoactive Drugs. 2013 Jan-Mar;45(1):28-38. doi: 10.1080/02791072.2013.763560. PMID 23662329
- [Background] Borges U, Pfannenstiel M, Tsukahara J, Laborde S, Klatt S, Raab M. Transcutaneous vagus nerve stimulation via tragus or cymba conchae: Are its psychophysiological effects dependent on the stimulation area? Int J Psychophysiol. 2021 Mar;161:64-75. doi: 10.1016/j.ijpsycho.2021.01.003. Epub 2021 Jan 11. PMID 33444689
- [Background] Brausch AM, Woods SE. Emotion Regulation Deficits and Nonsuicidal Self-Injury Prospectively Predict Suicide Ideation in Adolescents. Suicide Life Threat Behav. 2019 Jun;49(3):868-880. doi: 10.1111/sltb.12478. Epub 2018 Jun 14. PMID 29900570
- [Background] Brenner SL, Beauchaine TP. Pre-ejection period reactivity and psychiatric comorbidity prospectively predict substance use initiation among middle-schoolers: a pilot study. Psychophysiology. 2011 Nov;48(11):1588-1596. doi: 10.1111/j.1469-8986.2011.01230.x. Epub 2011 Jul 5. PMID 21729103
- [Background] Brent D. Nonsuicidal self-injury as a predictor of suicidal behavior in depressed adolescents. Am J Psychiatry. 2011 May;168(5):452-4. doi: 10.1176/appi.ajp.2011.11020215. No abstract available. PMID 21536697
- [Background] Brent DA, McMakin DL, Kennard BD, Goldstein TR, Mayes TL, Douaihy AB. Protecting adolescents from self-harm: a critical review of intervention studies. J Am Acad Child Adolesc Psychiatry. 2013 Dec;52(12):1260-71. doi: 10.1016/j.jaac.2013.09.009. Epub 2013 Sep 29. PMID 24290459
- [Background] Bresin K, Mekawi Y. Different Ways to Drown Out the Pain: A Meta-Analysis of the Association Between Nonsuicidal Self-Injury and Alcohol Use. Arch Suicide Res. 2022 Apr-Jun;26(2):348-369. doi: 10.1080/13811118.2020.1802378. Epub 2020 Aug 11. PMID 32780651
- [Background] Bretherton B, Atkinson L, Murray A, Clancy J, Deuchars S, Deuchars J. Effects of transcutaneous vagus nerve stimulation in individuals aged 55 years or above: potential benefits of daily stimulation. Aging (Albany NY). 2019 Jul 30;11(14):4836-4857. doi: 10.18632/aging.102074. PMID 31358702
- [Background] Burger AM, Van Diest I, Van der Does W, Korbee JN, Waziri N, Brosschot JF, Verkuil B. The effect of transcutaneous vagus nerve stimulation on fear generalization and subsequent fear extinction. Neurobiol Learn Mem. 2019 May;161:192-201. doi: 10.1016/j.nlm.2019.04.006. Epub 2019 Apr 12. PMID 30986531
- [Background] Burger AM, Van der Does W, Thayer JF, Brosschot JF, Verkuil B. Transcutaneous vagus nerve stimulation reduces spontaneous but not induced negative thought intrusions in high worriers. Biol Psychol. 2019 Mar;142:80-89. doi: 10.1016/j.biopsycho.2019.01.014. Epub 2019 Jan 30. PMID 30710565
- [Background] Centers for Disease Control. (2006). CDC injury fact book. Atlanta, GA: National Center for Injury Prevention Control.
- [Background] Centers for Disease Control (2020). Suicide rates in the United States continue to increase. Retrieved on 9/8/2020 from https://www.cdc.gov/nchs/products/databriefs/db309.htm#fig2
- [Background] Centers for Disease Control and Prevention (2021). Youth Risk Behavior Surveillance System (YRBSS) results. Downloaded on 6/22/2021 from https://www.cdc.gov/healthyyouth/data/yrbs/results.htm
- [Background] Clark DB, Thatcher DL, Martin CS. Child abuse and other traumatic experiences, alcohol use disorders, and health problems in adolescence and young adulthood. J Pediatr Psychol. 2010 Jun;35(5):499-510. doi: 10.1093/jpepsy/jsp117. Epub 2009 Dec 4. PMID 19966317
- [Background] ClinicalTrials.gov. (2021). A study of new treatment for excessive alcohol users by electric stimulation of nerves around the ear. Retrieved on 6/24/2021 from https://clinicaltrials.gov/ct2/show/NCT04106739
- [Background] Cohen JR, Thomsen KN, Tu KM, Thakur H, McNeil S, Menon SV. Cardiac autonomic functioning and post-traumatic stress: A preliminary study in youth at-risk for PTSD. Psychiatry Res. 2020 Feb;284:112684. doi: 10.1016/j.psychres.2019.112684. Epub 2019 Nov 7. PMID 31740215
- [Background] Cooper ML, Frone MR, Russell M, Mudar P. Drinking to regulate positive and negative emotions: a motivational model of alcohol use. J Pers Soc Psychol. 1995 Nov;69(5):990-1005. doi: 10.1037//0022-3514.69.5.990. PMID 7473043
- [Background] Crowell SE, Beauchaine TP, McCauley E, Smith CJ, Stevens AL, Sylvers P. Psychological, autonomic, and serotonergic correlates of parasuicide among adolescent girls. Dev Psychopathol. 2005 Fall;17(4):1105-27. doi: 10.1017/s0954579405050522. PMID 16613433
- [Background] Crowell SE, Beauchaine TP, McCauley E, Smith CJ, Vasilev CA, Stevens AL. Parent-child interactions, peripheral serotonin, and self-inflicted injury in adolescents. J Consult Clin Psychol. 2008 Feb;76(1):15-21. doi: 10.1037/0022-006X.76.1.15. PMID 18229978
- [Background] Crowell SE, Beauchaine TP, Linehan MM. A biosocial developmental model of borderline personality: Elaborating and extending Linehan's theory. Psychol Bull. 2009 May;135(3):495-510. doi: 10.1037/a0015616. PMID 19379027
- [Background] Crowell SE, Baucom BR, McCauley E, Potapova NV, Fitelson M, Barth H, Smith CJ, Beauchaine TP. Mechanisms of contextual risk for adolescent self-injury: invalidation and conflict escalation in mother-child interactions. J Clin Child Adolesc Psychol. 2013;42(4):467-80. doi: 10.1080/15374416.2013.785360. Epub 2013 Apr 14. PMID 23581508
- [Background] Crowell SE, Butner JE, Wiltshire TJ, Munion AK, Yaptangco M, Beauchaine TP. Evaluating Emotional and Biological Sensitivity to Maternal Behavior among Self-injuring and Depressed Adolescent Girls Using Nonlinear Dynamics. Clin Psychol Sci. 2017 Mar 1;5(2):272-285. doi: 10.1177/2167702617692861. Epub 2017 Mar 13. PMID 28924493
- [Background] Donovan JE, Molina BS. Childhood risk factors for early-onset drinking. J Stud Alcohol Drugs. 2011 Sep;72(5):741-51. doi: 10.15288/jsad.2011.72.741. PMID 21906502
- [Background] Dvorak RD, Sargent EM, Kilwein TM, Stevenson BL, Kuvaas NJ, Williams TJ. Alcohol use and alcohol-related consequences: associations with emotion regulation difficulties. Am J Drug Alcohol Abuse. 2014 Mar;40(2):125-30. doi: 10.3109/00952990.2013.877920. PMID 24588419
- [Background] Fang J, Rong P, Hong Y, Fan Y, Liu J, Wang H, Zhang G, Chen X, Shi S, Wang L, Liu R, Hwang J, Li Z, Tao J, Wang Y, Zhu B, Kong J. Transcutaneous Vagus Nerve Stimulation Modulates Default Mode Network in Major Depressive Disorder. Biol Psychiatry. 2016 Feb 15;79(4):266-73. doi: 10.1016/j.biopsych.2015.03.025. Epub 2015 Apr 2. PMID 25963932
- [Background] Fang J, Egorova N, Rong P, Liu J, Hong Y, Fan Y, Wang X, Wang H, Yu Y, Ma Y, Xu C, Li S, Zhao J, Luo M, Zhu B, Kong J. Early cortical biomarkers of longitudinal transcutaneous vagus nerve stimulation treatment success in depression. Neuroimage Clin. 2016 Dec 18;14:105-111. doi: 10.1016/j.nicl.2016.12.016. eCollection 2017. PMID 28180068
- [Background] Foley, J. O., & DuBois, F. S. (1937). Quantitative studies of the vagus nerve in the cat. I. The ratio of sensory to motor fibers. Journal of Comparative Neurology, 67, 49-67.
- [Background] Ford JD, Steinberg KL, Hawke J, Levine J, Zhang W. Randomized trial comparison of emotion regulation and relational psychotherapies for PTSD with girls involved in delinquency. J Clin Child Adolesc Psychol. 2012;41(1):27-37. doi: 10.1080/15374416.2012.632343. PMID 22233243
- [Background] Ford JD, Gomez JM. The relationship of psychological trauma and dissociative and posttraumatic stress disorders to nonsuicidal self-injury and suicidality: a review. J Trauma Dissociation. 2015;16(3):232-71. doi: 10.1080/15299732.2015.989563. Epub 2015 Mar 11. PMID 25758363
- [Background] Fox HC, Hong KA, Sinha R. Difficulties in emotion regulation and impulse control in recently abstinent alcoholics compared with social drinkers. Addict Behav. 2008 Feb;33(2):388-94. doi: 10.1016/j.addbeh.2007.10.002. Epub 2007 Oct 16. PMID 18023295
- [Background] Gadow, K. D., & Sprafkin, J. (2013). Child and Adolescent Symptom Inventory-5. Stony Brook, NY: Checkmate Plus.
- [Background] George MS, Rush AJ, Marangell LB, Sackeim HA, Brannan SK, Davis SM, Howland R, Kling MA, Moreno F, Rittberg B, Dunner D, Schwartz T, Carpenter L, Burke M, Ninan P, Goodnick P. A one-year comparison of vagus nerve stimulation with treatment as usual for treatment-resistant depression. Biol Psychiatry. 2005 Sep 1;58(5):364-73. doi: 10.1016/j.biopsych.2005.07.028. PMID 16139582
- [Background] Goldin PR, McRae K, Ramel W, Gross JJ. The neural bases of emotion regulation: reappraisal and suppression of negative emotion. Biol Psychiatry. 2008 Mar 15;63(6):577-86. doi: 10.1016/j.biopsych.2007.05.031. Epub 2007 Sep 21. PMID 17888411
- [Background] Graham JW. Missing data analysis: making it work in the real world. Annu Rev Psychol. 2009;60:549-76. doi: 10.1146/annurev.psych.58.110405.085530. PMID 18652544
- [Background] Gratz, K. L. & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54.
- [Background] Grossman P, van Beek J, Wientjes C. A comparison of three quantification methods for estimation of respiratory sinus arrhythmia. Psychophysiology. 1990 Nov;27(6):702-14. doi: 10.1111/j.1469-8986.1990.tb03198.x. PMID 2100356
- [Background] Haag K, Hiller R, Peyk P, Michael T, Meiser-Stedman R, Fearon P, Ehlers A, Halligan SL. A Longitudinal Examination of Heart-Rate and Heart Rate Variability as Risk Markers for Child Posttraumatic Stress Symptoms in an Acute Injury Sample. J Abnorm Child Psychol. 2019 Nov;47(11):1811-1820. doi: 10.1007/s10802-019-00553-2. PMID 31073881
- [Background] He W, Jing X, Wang X, Rong P, Li L, Shi H, Shang H, Wang Y, Zhang J, Zhu B. Transcutaneous auricular vagus nerve stimulation as a complementary therapy for pediatric epilepsy: a pilot trial. Epilepsy Behav. 2013 Sep;28(3):343-6. doi: 10.1016/j.yebeh.2013.02.001. Epub 2013 Jun 29. PMID 23820114
- [Background] Hewig, J., Hagemann, D., Seifert, J., Gollwitzer, M., Naumann, E., & Bartussek, D. (2005). A revised film set for the induction of basic emotions. Cognition and Emotion, 19(7), 1095-1109. doi:10.1080/ 02699930541000084
- [Background] Humeniuk R, Ali R, Babor TF, Farrell M, Formigoni ML, Jittiwutikarn J, de Lacerda RB, Ling W, Marsden J, Monteiro M, Nhiwatiwa S, Pal H, Poznyak V, Simon S. Validation of the Alcohol, Smoking And Substance Involvement Screening Test (ASSIST). Addiction. 2008 Jun;103(6):1039-47. doi: 10.1111/j.1360-0443.2007.02114.x. Epub 2008 Mar 28. PMID 18373724
- [Background] Hutcherson CA, Goldin PR, Ochsner KN, Gabrieli JD, Barrett LF, Gross JJ. Attention and emotion: does rating emotion alter neural responses to amusing and sad films? Neuroimage. 2005 Sep;27(3):656-68. doi: 10.1016/j.neuroimage.2005.04.028. PMID 15946863
- [Background] Johnson RL, Wilson CG. A review of vagus nerve stimulation as a therapeutic intervention. J Inflamm Res. 2018 May 16;11:203-213. doi: 10.2147/JIR.S163248. eCollection 2018. PMID 29844694
- [Background] Jongkees BJ, Immink MA, Finisguerra A, Colzato LS. Transcutaneous Vagus Nerve Stimulation (tVNS) Enhances Response Selection During Sequential Action. Front Psychol. 2018 Jul 6;9:1159. doi: 10.3389/fpsyg.2018.01159. eCollection 2018. PMID 30034357
- [Background] Kapetanovic, S., Gurdal, S., Ander, B., & Sorbring, E. (2021). Reported changes in adolescent psychosocial functioning during the COVID-19 outbreak. Adolescents, 1, 10-20. doi:10.3390/adolescents1010002
- [Background] Karpyak VM, Romanowicz M, Schmidt JE, Lewis KA, Bostwick JM. Characteristics of heart rate variability in alcohol-dependent subjects and nondependent chronic alcohol users. Alcohol Clin Exp Res. 2014 Jan;38(1):9-26. doi: 10.1111/acer.12270. Epub 2013 Oct 11. PMID 24117482
- [Background] Klonsky ED. The functions of deliberate self-injury: a review of the evidence. Clin Psychol Rev. 2007 Mar;27(2):226-39. doi: 10.1016/j.cpr.2006.08.002. Epub 2006 Oct 2. PMID 17014942
- [Background] Klonsky ED. The functions of self-injury in young adults who cut themselves: clarifying the evidence for affect-regulation. Psychiatry Res. 2009 Apr 30;166(2-3):260-8. doi: 10.1016/j.psychres.2008.02.008. Epub 2009 Mar 10. PMID 19275962
- [Background] Klonsky ED, Glenn CR, Styer DM, Olino TM, Washburn JJ. The functions of nonsuicidal self-injury: converging evidence for a two-factor structure. Child Adolesc Psychiatry Ment Health. 2015 Sep 28;9:44. doi: 10.1186/s13034-015-0073-4. eCollection 2015. PMID 26421059
- [Background] Koenig J, Parzer P, Haigis N, Liebemann J, Jung T, Resch F, Kaess M. Effects of acute transcutaneous vagus nerve stimulation on emotion recognition in adolescent depression. Psychol Med. 2021 Feb;51(3):511-520. doi: 10.1017/S0033291719003490. Epub 2019 Dec 10. PMID 31818339
- [Background] Kong J, Fang J, Park J, Li S, Rong P. Treating Depression with Transcutaneous Auricular Vagus Nerve Stimulation: State of the Art and Future Perspectives. Front Psychiatry. 2018 Feb 5;9:20. doi: 10.3389/fpsyt.2018.00020. eCollection 2018. PMID 29459836
- [Background] Kuntsche E, Knibbe R, Gmel G, Engels R. Why do young people drink? A review of drinking motives. Clin Psychol Rev. 2005 Nov;25(7):841-61. doi: 10.1016/j.cpr.2005.06.002. PMID 16095785
- [Background] Linehan, M. M., & Comtois, K. A. (1996). Lifetime parasuicide count: Unpublished manuscript.
- [Background] Linehan, M. M., Comtois, K. A., & Ward-Ciesielski, E. F. (2012). Assessing and managing risk with suicidal individuals. Cognitive and Behavioral Practice,19(2), 218-232.
- [Background] Linehan, M. M. (2014). DBT training manual. New York, NY: Guilford Press.
- [Background] Linehan, M. M. (2015). DBT skills training handouts and worksheets. New York, NY: Guilford.
- [Background] Liu J, Fang J, Wang Z, Rong P, Hong Y, Fan Y, Wang X, Park J, Jin Y, Liu C, Zhu B, Kong J. Transcutaneous vagus nerve stimulation modulates amygdala functional connectivity in patients with depression. J Affect Disord. 2016 Nov 15;205:319-326. doi: 10.1016/j.jad.2016.08.003. Epub 2016 Aug 11. PMID 27559632
- [Background] Marangell LB, Rush AJ, George MS, Sackeim HA, Johnson CR, Husain MM, Nahas Z, Lisanby SH. Vagus nerve stimulation (VNS) for major depressive episodes: one year outcomes. Biol Psychiatry. 2002 Feb 15;51(4):280-7. doi: 10.1016/s0006-3223(01)01343-9. PMID 11958778
- [Background] McDonough-Caplan H, Klein DN, Beauchaine TP. Comorbidity and continuity of depression and conduct problems from elementary school to adolescence. J Abnorm Psychol. 2018 Apr;127(3):326-337. doi: 10.1037/abn0000339. Epub 2018 Feb 26. PMID 29481099
- [Background] Miller JC, Horvath SM. Impedance cardiography. Psychophysiology. 1978 Jan;15(1):80-91. doi: 10.1111/j.1469-8986.1978.tb01340.x. No abstract available. PMID 625525
- [Background] Moran P, Coffey C, Romaniuk H, Degenhardt L, Borschmann R, Patton GC. Substance use in adulthood following adolescent self-harm: a population-based cohort study. Acta Psychiatr Scand. 2015 Jan;131(1):61-8. doi: 10.1111/acps.12306. Epub 2014 Jun 23. PMID 24954250
- [Background] Muller HHO, Moeller S, Lucke C, Lam AP, Braun N, Philipsen A. Vagus Nerve Stimulation (VNS) and Other Augmentation Strategies for Therapy-Resistant Depression (TRD): Review of the Evidence and Clinical Advice for Use. Front Neurosci. 2018 Apr 10;12:239. doi: 10.3389/fnins.2018.00239. eCollection 2018. PMID 29692707
- [Background] National Institute of Mental Health. (2021). NIMH Strategic Plan for Research. Retrieved on 6/21/2021 from https://iamhrf.org/sites/iamhrf.org/files/uploads/publication/files/nimh_strategicplanforresearch.pdf
- [Background] National Institute on Alcohol Abuse and Alcoholism. (2021). NIAAA Strategic Plan. Downloaded on 6/21/2021 from https://www.niaaa.nih.gov/strategic-plan.
- [Background] Neumann A, van Lier PA, Gratz KL, Koot HM. Multidimensional assessment of emotion regulation difficulties in adolescents using the Difficulties in Emotion Regulation Scale. Assessment. 2010 Mar;17(1):138-49. doi: 10.1177/1073191109349579. Epub 2009 Nov 14. PMID 19915198
- [Background] Neuvana(a). (2021). Xen. Retrieved on 6/27/2021 from https://neuvanalife.com/products/xen
- [Background] Neuvana(b). (2021). Neuvana. Retrieved on 8/24/2021 from https://neuvanalife.com/
- [Background] McManama O'Brien KH, Becker SJ, Spirito A, Simon V, Prinstein MJ. Differentiating adolescent suicide attempters from ideators: examining the interaction between depression severity and alcohol use. Suicide Life Threat Behav. 2014 Feb;44(1):23-33. doi: 10.1111/sltb.12050. Epub 2013 Jul 25. PMID 23889515
- [Background] Oetzel, B. K., & Scherer, D. G. (2003). Therapeutic engagement with adolescents in psychotherapy. Psychotherapy: Theory, Research, Practice, Training, 40, 215-225. doi:10.1037/0033-3204.40.3.215
- [Background] O'Reardon JP, Cristancho P, Peshek AD. Vagus Nerve Stimulation (VNS) and Treatment of Depression: To the Brainstem and Beyond. Psychiatry (Edgmont). 2006 May;3(5):54-63. PMID 21103178
- [Background] Patrick ME, Schulenberg JE, O'Malley PM, Johnston LD, Bachman JG. Adolescents' reported reasons for alcohol and marijuana use as predictors of substance use and problems in adulthood. J Stud Alcohol Drugs. 2011 Jan;72(1):106-16. doi: 10.15288/jsad.2011.72.106. PMID 21138717
- [Background] Penry JK, Dean JC. Prevention of intractable partial seizures by intermittent vagal stimulation in humans: preliminary results. Epilepsia. 1990;31 Suppl 2:S40-3. doi: 10.1111/j.1528-1157.1990.tb05848.x. PMID 2121469
- [Background] Perepletchikova F, Nathanson D, Axelrod SR, Merrill C, Walker A, Grossman M, Rebeta J, Scahill L, Kaufman J, Flye B, Mauer E, Walkup J. Randomized Clinical Trial of Dialectical Behavior Therapy for Preadolescent Children With Disruptive Mood Dysregulation Disorder: Feasibility and Outcomes. J Am Acad Child Adolesc Psychiatry. 2017 Oct;56(10):832-840. doi: 10.1016/j.jaac.2017.07.789. Epub 2017 Aug 10. PMID 28942805
- [Background] Porges SW. Orienting in a defensive world: mammalian modifications of our evolutionary heritage. A Polyvagal Theory. Psychophysiology. 1995 Jul;32(4):301-18. doi: 10.1111/j.1469-8986.1995.tb01213.x. PMID 7652107
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Prechtl JC, Powley TL. The fiber composition of the abdominal vagus of the rat. Anat Embryol (Berl). 1990;181(2):101-15. doi: 10.1007/BF00198950. PMID 2327594
- [Background] Quintana DS, McGregor IS, Guastella AJ, Malhi GS, Kemp AH. A meta-analysis on the impact of alcohol dependence on short-term resting-state heart rate variability: implications for cardiovascular risk. Alcohol Clin Exp Res. 2013 Jan;37 Suppl 1:E23-9. doi: 10.1111/j.1530-0277.2012.01913.x. Epub 2012 Jul 26. PMID 22834996
- [Background] Rathus, J. H., & Miller, A. L. (2014). DBT Skills Manual for adolescents. New York: Guilford Press.
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648
- [Background] Reynolds, W. M. (1987). Suicidal Ideation Questionnaire-Junior. Odessa, FL: Psychological Assessment Resources.
- [Background] Reynolds, W. M. (1988). Suicidal Ideation Questionnaire: Professional manual. Odessa, FL: Psychological Assessment Resources.
- [Background] Reynolds SK, Lindenboim N, Comtois KA, Murray A, Linehan MM. Risky assessments: participant suicidality and distress associated with research assessments in a treatment study of suicidal behavior. Suicide Life Threat Behav. 2006 Feb;36(1):19-34. doi: 10.1521/suli.2006.36.1.19. PMID 16676622
- [Background] Rong PJ, Fang JL, Wang LP, Meng H, Liu J, Ma YG, Ben H, Li L, Liu RP, Huang ZX, Zhao YF, Li X, Zhu B, Kong J. Transcutaneous vagus nerve stimulation for the treatment of depression: a study protocol for a double blinded randomized clinical trial. BMC Complement Altern Med. 2012 Dec 14;12:255. doi: 10.1186/1472-6882-12-255. PMID 23241431
- [Background] Rong P, Liu J, Wang L, Liu R, Fang J, Zhao J, Zhao Y, Wang H, Vangel M, Sun S, Ben H, Park J, Li S, Meng H, Zhu B, Kong J. Effect of transcutaneous auricular vagus nerve stimulation on major depressive disorder: A nonrandomized controlled pilot study. J Affect Disord. 2016 May;195:172-9. doi: 10.1016/j.jad.2016.02.031. Epub 2016 Feb 10. PMID 26896810
- [Background] Sauder CL, Derbidge CM, Beauchaine TP. Neural responses to monetary incentives among self-injuring adolescent girls. Dev Psychopathol. 2016 Feb;28(1):277-91. doi: 10.1017/S0954579415000449. Epub 2015 Jun 8. PMID 26050788
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Sayette MA. The effects of alcohol on emotion in social drinkers. Behav Res Ther. 2017 Jan;88:76-89. doi: 10.1016/j.brat.2016.06.005. PMID 28110679
- [Background] Schmitz WM Jr, Allen MH, Feldman BN, Gutin NJ, Jahn DR, Kleespies PM, Quinnett P, Simpson S. Preventing suicide through improved training in suicide risk assessment and care: an American Association of Suicidology Task Force report addressing serious gaps in U.S. mental health training. Suicide Life Threat Behav. 2012 Jun;42(3):292-304. doi: 10.1111/j.1943-278X.2012.00090.x. Epub 2012 Apr 11. PMID 22494118
- [Background] Naeger S. Emergency Department Visits Involving Underage Alcohol Misuse: 2010 to 2013. 2017 May 16. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK436366/ PMID 28632359
- [Background] Swannell SV, Martin GE, Page A, Hasking P, St John NJ. Prevalence of nonsuicidal self-injury in nonclinical samples: systematic review, meta-analysis and meta-regression. Suicide Life Threat Behav. 2014 Jun;44(3):273-303. doi: 10.1111/sltb.12070. Epub 2014 Jan 15. PMID 24422986
- [Background] Thayer JF, Lane RD. Claude Bernard and the heart-brain connection: further elaboration of a model of neurovisceral integration. Neurosci Biobehav Rev. 2009 Feb;33(2):81-8. doi: 10.1016/j.neubiorev.2008.08.004. Epub 2008 Aug 13. PMID 18771686
- [Background] Tuisku V, Kiviruusu O, Pelkonen M, Karlsson L, Strandholm T, Marttunen M. Depressed adolescents as young adults - predictors of suicide attempt and non-suicidal self-injury during an 8-year follow-up. J Affect Disord. 2014 Jan;152-154:313-9. doi: 10.1016/j.jad.2013.09.031. Epub 2013 Oct 5. PMID 24144580
- [Background] UL. (2021). Certification. Retrieved on 8/24/2021 from https://www.ul.com/services/certification
- [Background] Valentine SE, Bankoff SM, Poulin RM, Reidler EB, Pantalone DW. The use of dialectical behavior therapy skills training as stand-alone treatment: a systematic review of the treatment outcome literature. J Clin Psychol. 2015 Jan;71(1):1-20. doi: 10.1002/jclp.22114. Epub 2014 Jul 14. PMID 25042066
- [Background] van den Bosch LM, Verheul R, Schippers GM, van den Brink W. Dialectical Behavior Therapy of borderline patients with and without substance use problems. Implementation and long-term effects. Addict Behav. 2002 Nov-Dec;27(6):911-23. doi: 10.1016/s0306-4603(02)00293-9. PMID 12369475
- [Background] Verma N, Mudge JD, Kasole M, Chen RC, Blanz SL, Trevathan JK, Lovett EG, Williams JC, Ludwig KA. Auricular Vagus Neuromodulation-A Systematic Review on Quality of Evidence and Clinical Effects. Front Neurosci. 2021 Apr 30;15:664740. doi: 10.3389/fnins.2021.664740. eCollection 2021. PMID 33994937
- [Background] Wang Z, Fang J, Liu J, Rong P, Jorgenson K, Park J, Lang C, Hong Y, Zhu B, Kong J. Frequency-dependent functional connectivity of the nucleus accumbens during continuous transcutaneous vagus nerve stimulation in major depressive disorder. J Psychiatr Res. 2018 Jul;102:123-131. doi: 10.1016/j.jpsychires.2017.12.018. Epub 2017 Dec 28. PMID 29674268
- [Background] Weissman DG, Bitran D, Miller AB, Schaefer JD, Sheridan MA, McLaughlin KA. Difficulties with emotion regulation as a transdiagnostic mechanism linking child maltreatment with the emergence of psychopathology. Dev Psychopathol. 2019 Aug;31(3):899-915. doi: 10.1017/S0954579419000348. Epub 2019 Apr 8. PMID 30957738
- [Background] Williams F, Hasking P. Emotion regulation, coping and alcohol use as moderators in the relationship between non-suicidal self-injury and psychological distress. Prev Sci. 2010 Mar;11(1):33-41. doi: 10.1007/s11121-009-0147-8. PMID 19707873
- [Background] Wittbrodt MT, Gurel NZ, Nye JA, Ladd S, Shandhi MMH, Huang M, Shah AJ, Pearce BD, Alam ZS, Rapaport MH, Murrah N, Ko YA, Haffer AA, Shallenberger LH, Vaccarino V, Inan OT, Bremner JD. Non-invasive vagal nerve stimulation decreases brain activity during trauma scripts. Brain Stimul. 2020 Sep-Oct;13(5):1333-1348. doi: 10.1016/j.brs.2020.07.002. Epub 2020 Jul 10. PMID 32659483
- [Background] Wolff JC, Thompson E, Thomas SA, Nesi J, Bettis AH, Ransford B, Scopelliti K, Frazier EA, Liu RT. Emotion dysregulation and non-suicidal self-injury: A systematic review and meta-analysis. Eur Psychiatry. 2019 Jun;59:25-36. doi: 10.1016/j.eurpsy.2019.03.004. Epub 2019 Apr 12. PMID 30986729
- [Background] Zalewski M, Lewis JK, Martin CG. Identifying novel applications of dialectical behavior therapy: considering emotion regulation and parenting. Curr Opin Psychol. 2018 Jun;21:122-126. doi: 10.1016/j.copsyc.2018.02.013. Epub 2018 Mar 1. PMID 29529427